CLINICAL TRIAL: NCT03023163
Title: A Longitudinal Examination of Aging With a Spinal Cord Injury: Cardiovascular, Cerebrovascular and Cognitive Consequences
Status: Completed | Type: Observational
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Research Health Scientist, James J. Peters Veterans Affairs Medical Center
Other Study IDs: WEC-16-039
Record Dates: First submitted 2016-12-27; First posted 2017-01-18 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Spinal Cord Injury
Keywords: autonomic dysreflexia; baroreceptor integrity; sympathetic integrity; vagal integrity; autonomic integrity; arterial stiffness; cognitive function; traumatic brain injury; cerebral blood flow; white matter hyperintensities; cerebral vascular resistance index
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Older SCI: Individuals that are between the ages of 50-75 years old, have a traumatic SCI, level of injury between C1-T12, non-ambulatory (wheelchair dependent), AIS grade A, B, or C, and injury occurred more than 1 year ago.
- Older Able-Bodied Controls: Individuals that are between the ages of 50-75 years old and primary language is English.
- Longitudinal SCI: Individuals that are between the ages of 28-54 years old and previously participated in the Impact of Age on Cardiovascular, Cerebrovascular, and Cognitive Health study in a 3-5 year span.
  Interventions: Other: Longitudinal
- Longitudinal Able-Bodied Controls: Individuals that are between the ages of 28-54 years old and previously participated in the Impact of Age on Cardiovascular, Cerebrovascular, and Cognitive Health study in a 3-5 year span.
  Interventions: Other: Longitudinal

INTERVENTIONS:
Other: Longitudinal — Participants that completed the Impact of Age on Cardiovascular, Cerebrovascular, Cerebrovascular and Cognitive Health study, will be re-assessed again to compare longitudinal (3-5 years) change in blood pressure, cerebral blood flow, arterial stiffness and cognitive health.
  Groups: Longitudinal Able-Bodied Controls; Longitudinal SCI

SUMMARY:
The general population is aging, today 12% of the United States population is older than 65 and it is estimated that by 2020 the number of people in the United States older than 65 will outnumber children younger than 5. As the general population ages, the spinal cord injury (SCI) population is also aging and it is estimated that 14% is older than 60. Although persons with SCI are living longer, life expectancy remains below that of the general population with cardiovascular and cerebrovascular diseases accounting for more than 25% of all deaths since 1995. Similar to findings in the general population, BP dysregulation may impact cognitive function, and investigators reported poorer performance on tasks of memory and attention processing in hypotensive individuals with SCI compared to a normotensive SCI cohort. Thus, it is imperative that investigators work to minimize the impact of cognitive deficits on these aspects of life quality in persons with SCI as they age. Therefore the goals of this study are: Study 1) to compare cardiovascular, cerebrovascular and cognitive function and fMRI between older individuals with SCI (50-75 years) and older age-matched controls and Study 2) to determine 3-5 year longitudinal changes in cardiovascular, cerebrovascular and cognitive function and fMRI in relatively young individuals with SCI (28-54 years) compared to relatively young age-matched controls.

DETAILED DESCRIPTION:
All potential subjects will undergo a two-part screening process which consists of an initial screening via telephone and a detailed, in-person screening. Eligible subjects will be invited to participate in a 4 hour laboratory visit during which their arterial stiffness, blood pressure, heart rate, respiration rate and, blood flow to the brain will be monitored at rest and during a comprehensive series of cognitive tests. For Study 1 (cross-sectional), 40 older (50-75 years) individuals with SCI and 20 age-matched non-SCI controls will be recruited. For study 2 (longitudinal), 30 individuals (28-54 years) with SCI and 20 age-matched non-SCI will be recruited from previous enrollment in the Impact of Age on Cardiovascular, Cerebrovascular and Cognitive Health in SCI study to learn the longitudinal changes in cardiovascular, cerebrovascular and cognitive health.

ELIGIBILITY:
Inclusion Criteria:

* Study 1) Between the ages of 50-75 years old
* Study 2) Between the ages of 28-54 years old
* Completed Impact of Age on Cardiovascular, Cerebrovascular and Cognitive Health study
* For Both:
* Primary language is English
* Additional Inclusion Criteria: SCI Subjects
* Level of injury between C1-T12;
* Non-ambulatory (wheelchair dependent);
* AIS grade A, B, or C;
* Injury occurred more than 1 year ago.

Exclusion Criteria:

* Acute illness or infection;
* Controlled or uncontrolled hypertension or Diabetes mellitus;
* Documented history of traumatic brain injury;
* Stroke
* Epilepsy or seizure disorders;
* Multiple sclerosis & Parkinson's disease;
* Psychiatric disorders (post-traumatic stress disorder, schizophrenia, bipolar disorder);
* Alzheimer's disease & dementia

Ages: 28 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study 1) 40 older (50-75 years) individuals with SCI and 20 age-matched non-SCI controls.
  Study 2) 30 individuals (28-54 years) with SCI and 20 age-matched non-SCI controls. Participants will be recruited from the Impact of Age on Cardiovascular, Cerebrovascular and Cognitive Health study.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure (mmHg) | Up to 3 years
  To determine change in systolic blood pressure from seated rest to seated cognitive testing in subjects with and without spinal cord injury.

SECONDARY OUTCOMES:
Performance on tests of memory (PASAT) and processing speed (SDMT). | Up to 3 years
  To compere cognitive performance on tests of working memory and processing speed in individuals with and without spinal cord injury.
Cerebral Blood Flow Velocity (cm/second) from the middle cerebral arteries | Up to 3 years
  To determine change in cerebral blood flow velocity from seated rest to seated cognitive testing in subjects with and without spinal cord injury.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Wecht, EdD, Principal Investigator — James J Peters VA Medical Center
Locations (1):
- Kessler Foundation Research Center, West Orange, New Jersey, United States